CLINICAL TRIAL: NCT04866862
Title: A Single Arm, Open Label, Phase II, Exploratory Study of Fruquitinib Combined With Camrelizumab in Non MSI-H / dMMR Refractory Colorectal Cancer.
Brief Title: Fruquitinib Combined With Camrelizumab in Non MSI-H/dMMR Refractory Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KEEP-G 05
Record Dates: First submitted 2021-03-28; First posted 2021-04-30 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Colorectal Neoplasm
Keywords: colorectal cancer; non MSI-H/dMMR; Camrelizumab; Fruquintinib
MeSH Terms: conditions — Colorectal Neoplasms | interventions — camrelizumab; HMPL-013

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combination of Fruquintinib and Camrelizumab (Experimental): Fruquintinib 5mg d1-21+ Camrelizumab 200mg d1; Repeated every 4 weeks
  Interventions: Drug: Combination of Fruquintinib and Camrelizumab

INTERVENTIONS:
Drug: Combination of Fruquintinib and Camrelizumab — Fruquintinib 5mg d1-21+Camrelizumab 200 mg d1
  Other Names: Fruquintinib 5mg d1-21+Camrelizumab 200 mg d1

SUMMARY:
Limited agents are optional after standard first and second line treatment for mCRC. Nowadays, cancer therapy has entered the era of immunotherapy. The approved cancer therapies include pembrolizumab and nivolumab, but only for MSI-H patients. 95% of non MSI-H / dMMR patients with advanced colorectal cancer can not benefit from them. Therefore, the use of PD-1 / PD-L1 monoclonal antibody in mCRC is greatly limited. Our previous research showed that anti-PD-1 combined with Fruquintinib can significantly inhibit the growth of CRC in MSS mice. At the same time, a retrospective clinical study showed that patients with MSS CRC can benefit from Sintilimab combined with Fruquintinib. Camrelizumab is PD-1 monoclonal antibody, which has been approved for a variety of tumors. The prospective clinical trial of Camrelizumab combined with Fruquintinib may bring new hope for the treatment of non MSI-H / dMMR patients with mCRC.This study is aimed to explore the efficacy, safety in advanced colorectal cancer failed to standard therapy in Chinese population.

DETAILED DESCRIPTION:
Our previous research showed that anti-PD-1 combined with Fruquintinib can significantly inhibit the growth of CRC in MSS mice. At the same time, a retrospective clinical study showed that patients with MSS CRC can benefit from Sintilimab combined with Fruquintinib. Camrelizumab is PD-1 monoclonal antibody, which has been approved for a variety of tumors. The prospective clinical trial of Camrelizumab combined with Fruquintinib may bring new hope for the treatment of non MSI-H / dMMR patients with mCRC.This study is aimed to explore the efficacy, safety in advanced colorectal cancer failed to standard therapy in Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological documentation of adenocarcinoma of the colon or rectum. All other histological types are excluded.
* Subjects with non MSI-H / dMMR metastatic colorectal cancer(CRC) (Stage IV)
* Subjects must have failed at least two lines of prior treatment, which must include a fluoropyrimidine, oxaliplatin and irinotecan.
* Subjects must not have been treated with Fruquitinib or any anti-PD-1 inhibitors.
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria, version 1.1.is necessary.
* Adequate bone marrow, liver, cardiac and renal function as assessed by the laboratory required by protocol.
* Assigned informed consent.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
* Life expectancy of at least 3 months.
* Subjects must complete the treatment and follow-up on schedule according to the research plan.
* No brain metastasis, no spinal cord compression.
* Subjects agree to use blood samples for study analysis.
* Women of childbearing age must be negative in pregnancy test and willing to take effective contraceptive measures during the study period.

Exclusion Criteria:

* Subjects are severe malnutrition or need tube feeding.
* Radiotherapy or surgery has been performed within 30 days before treatment.
* Previous treatment with anti-PD-1 / PD-L1 inhibitor and / or fruquitinib.
* Other malignant tumors within 2 years and without cure (except for cured basal cell carcinoma of skin and carcinoma in situ of cervix);
* Subjects have active autoimmune system diseases、systemic hormone therapy or anti autoimmune drug therapy.
* Subjects with immunodeficiency or receiving systemic steroid therapy (prednisone > 10 mg / day or other equivalent drugs) or other forms of immunosuppressive therapy 7 days before the first dose of combination therapy in this study;
* Subjects with active infection and still need systemic treatment 7 days before the first dose of therapy in this study.
* Subjects with uncontrollable systemic diabetes.
* Subjects with interstitial lung disease, non infectious pneumonia or pulmonary fibrosis;
* Subjects who have received allogeneic organ or stem cell transplantation in the past.
* Subjects allergic to the drugs or related components involved in this study.
* Are participating in other interventional clinical studies.
* The previous anti-tumor related adverses do not return to grade 1 in CTCAE before the first combination therapy.
* Subjects who have uncontrolled hypertension by drugs, that is, systolic blood pressure ≥ 140 mmHg and / or diastolic blood pressure ≥ 90 mmHg.
* Thrombotic or hemorrhagic tendency or history within 60 days before the first medication, regardless of the severity.
* Any serious or unstable medical condition、mental illness or known active alcohol or drug abuse or dependence.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-04-26 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | up to 2 years
  The percentage of subjects with total number of Complete Response (CR) + total number of Partial Response (PR)

SECONDARY OUTCOMES:
Progression-free Survival(PFS) | From date of subjects until the date of first documented progression or death from any cause, whichever came first, assessed up to 24 months
  PFS was defined as the time from assignment to disease progression radiological/clinical or death due to any cause, whichever occurs first. Subjects without progression or death at the time of analysis were censored at their last date of tumor evaluation.
Overall Survival (OS) | From assignment of the first subject until 32 death events observed, up to 2 years.
  OS is defined as the time from date of assignment to death due to any cause. Subjects still alive at the time of analysis were censored at their last date of last contact.
Disease control rate (DCR) | up to 2 years
  DCR is defined as the percentage of subjects whose best response was not Progressive Disease (PD) according to Response Evaluation Criteria in Solid Tumors (RECIST) (= total number of Complete Response (CR) + total number of Partial Response (PR) + total number of Stable Disease (SD)
Tumor Mutation Burden (TMB) | up to 2 years
  The total number of somatic gene coding error, base substitution. gene insertions or deletions in every million base detected.

OTHER OUTCOMES:
immunocytes and cell factor | up to 2 years
  The concentration of immunocytes and cell factor in the blood of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Wang, Study Chair — the first affilated hospital with Nanjing Medical University
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jacquelot N, Yamazaki T, Roberti MP, Duong CPM, Andrews MC, Verlingue L, Ferrere G, Becharef S, Vetizou M, Daillere R, Messaoudene M, Enot DP, Stoll G, Ugel S, Marigo I, Foong Ngiow S, Marabelle A, Prevost-Blondel A, Gaudreau PO, Gopalakrishnan V, Eggermont AM, Opolon P, Klein C, Madonna G, Ascierto PA, Sucker A, Schadendorf D, Smyth MJ, Soria JC, Kroemer G, Bronte V, Wargo J, Zitvogel L. Sustained Type I interferon signaling as a mechanism of resistance to PD-1 blockade. Cell Res. 2019 Oct;29(10):846-861. doi: 10.1038/s41422-019-0224-x. Epub 2019 Sep 3. PMID 31481761
- [Result] Brahmer JR, Drake CG, Wollner I, Powderly JD, Picus J, Sharfman WH, Stankevich E, Pons A, Salay TM, McMiller TL, Gilson MM, Wang C, Selby M, Taube JM, Anders R, Chen L, Korman AJ, Pardoll DM, Lowy I, Topalian SL. Phase I study of single-agent anti-programmed death-1 (MDX-1106) in refractory solid tumors: safety, clinical activity, pharmacodynamics, and immunologic correlates. J Clin Oncol. 2010 Jul 1;28(19):3167-75. doi: 10.1200/JCO.2009.26.7609. Epub 2010 Jun 1. PMID 20516446
- [Result] Le DT, Durham JN, Smith KN, Wang H, Bartlett BR, Aulakh LK, Lu S, Kemberling H, Wilt C, Luber BS, Wong F, Azad NS, Rucki AA, Laheru D, Donehower R, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Greten TF, Duffy AG, Ciombor KK, Eyring AD, Lam BH, Joe A, Kang SP, Holdhoff M, Danilova L, Cope L, Meyer C, Zhou S, Goldberg RM, Armstrong DK, Bever KM, Fader AN, Taube J, Housseau F, Spetzler D, Xiao N, Pardoll DM, Papadopoulos N, Kinzler KW, Eshleman JR, Vogelstein B, Anders RA, Diaz LA Jr. Mismatch repair deficiency predicts response of solid tumors to PD-1 blockade. Science. 2017 Jul 28;357(6349):409-413. doi: 10.1126/science.aan6733. Epub 2017 Jun 8. PMID 28596308
- [Result] Xu J, Zhang Y, Jia R, Yue C, Chang L, Liu R, Zhang G, Zhao C, Zhang Y, Chen C, Wang Y, Yi X, Hu Z, Zou J, Wang Q. Anti-PD-1 Antibody SHR-1210 Combined with Apatinib for Advanced Hepatocellular Carcinoma, Gastric, or Esophagogastric Junction Cancer: An Open-label, Dose Escalation and Expansion Study. Clin Cancer Res. 2019 Jan 15;25(2):515-523. doi: 10.1158/1078-0432.CCR-18-2484. Epub 2018 Oct 22. PMID 30348638
- [Result] Mei Q, Zhang W, Liu Y, Yang Q, Rasko JEJ, Nie J, Liu J, Li X, Dong L, Chen M, Zhang Y, Shi L, Wu H, Han W. Camrelizumab Plus Gemcitabine, Vinorelbine, and Pegylated Liposomal Doxorubicin in Relapsed/Refractory Primary Mediastinal B-Cell Lymphoma: A Single-Arm, Open-Label, Phase II Trial. Clin Cancer Res. 2020 Sep 1;26(17):4521-4530. doi: 10.1158/1078-0432.CCR-20-0514. Epub 2020 Jun 4. PMID 32499235
- [Result] Shirley M. Fruquintinib: First Global Approval. Drugs. 2018 Nov;78(16):1757-1761. doi: 10.1007/s40265-018-0998-z. PMID 30357594